CLINICAL TRIAL: NCT05522699
Title: Cough Suppressive Therapy in Chronic Cough: Randomized Controlled Trial
Brief Title: Cough Suppressive Therapy in Patients With Chronic Cough
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 974599
Record Dates: First submitted 2022-08-22; First posted 2022-08-31 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cough suppressive therapy (Experimental): The cough suppressive therapy consists of four one-to-one treatment sessions, 45 minutes per session, over a 2 months period. The sessions include patient education about chronic cough; negative effects of repeated cough as well as patient education of voluntary control of cough; identification of cough triggers and learning cough suppression techniques, and psychoeducational counselling including patient self-motivation, repetition of aims and techniques, behavior modification regarding over-awareness of the need to cough.
  The sessions will be conducted by a specially trained physiotherapist or speech and language therapist. All components of the cough suppressive therapy will be delivered to each participant but the focus and emphasis on individual techniques will be individually tailored for each participant, determined by the physio- or speech and language therapist together with the participant.
  Interventions: Behavioral: Cough suppressive therapy
- Healthy lifestyle instructions (Active Comparator): The Healthy lifestyle instructions consists of four one-to-one treatment sessions, 30 minutes per session, over a 2 months period. The sessions will be conducted by a specially trained physiotherapist or speech and language therapist. The sessions include patient education and motivational conversation about healthy eating habits, physical activity, stress and relaxation.
  Interventions: Behavioral: General healthy lifestyle instructions

INTERVENTIONS:
Behavioral: Cough suppressive therapy — The cough suppressive therapy based on the treatment regime "Physiotherapy, and speech and language therapy intervention for patients with refractory chronic cough (PSALTI) developed by S. Chamberlain et al (Thorax. 2017 Feb;72(2):129-136).
  Arms: Cough suppressive therapy
Behavioral: General healthy lifestyle instructions — The general healthy lifestyle instructions are based on the recommendations from the The Public Health Agency of Sweden.
  Arms: Healthy lifestyle instructions

SUMMARY:
In this randomized, placebo-controlled, interventional study on chronic cough a non-pharmacological cough suppressive therapy is the intervention to be studied, with a control group receiving treatment consisting of general healthy lifestyle advice. The following data will be collected before, after and up to six months after treatment: Standardized questionnaires for diagnosis of background factors, Leicester Cough Questionnaire (LCQ), Work Ability Index (WAI), and cough frequency as well as lung function and biomarkers.

The primary treatment effect measurement will be changes in chronic cough-related quality of life, measured by the Leicester Cough Questionnaire (LCQ).

DETAILED DESCRIPTION:
The study will be carried out in collaboration between respiratory physicians, clinical physiologists, physiotherapists, speech- and language therapists and gastroenterologists.

The primary hypothesis of the planned study is:

The cough suppressive therapy improves chronic cough-related quality of life and work ability, and is sustained over six months after treatment.

The secondary hypotheses of the planned study are:

Treatment of chronic cough by the cough suppressive therapy can reduce cough frequency (measured by an automated cough detector), airway inflammation and airway resistance.

Baseline differences in clinical findings, biomarkers and physiologic measurements predict different treatment effects.

The following data will be collected before and after treatment:

* Standardized questionnaires for diagnosis of background factors and cough duration, LCQ, WAI, questions on sick leave days, voice disturbance questionnaire.
* Physiological measurements: Spirometry with reversibility test, impulse oscillometry before and after provocation with hypertonic saline inhalation. 24 hours cough frequency analysis, voice analysis.
* Biomarkers: Fractional exhaled nitric oxide (FeNO), blood-eosinophils and eosinophil cationic protein in serum, proteomics in particles in exhaled air (PExA)

ELIGIBILITY:
Inclusion Criteria:

* Chronic cough (duration >2 months) without a structural lung disease and a normal chest X-ray, which have failed pharmacological treatment.
* Being able to understand the swedish language.

Exclusion Criteria:

* Pulmonary abnormalities on a chest X-ray, structural lung disease, or chronic obstructive pulmonary disease (COPD) of spirometry stage Global Initiative for Obstructive Lung Disease (GOLD) 2 or higher.
* Smoking under the last three months.
* Ongoing or recent treatment with angiotensin-converting enzyme (ACE) inhibitor
* Active aspiration, vocal cord nodules or upper respiratory tract infection in the previous 4 weeks.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-03 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Leicester Cough Questionnaire (LCQ) | Change from baseline LCQ at one week and 6 months after completed intervention
  Leicester Cough Questionnaire (LCQ) is an English-born self-reporting quality of life measure of chronic cough,

SECONDARY OUTCOMES:
Change in The Work Ability Index (WAI) | Change from baseline WAI at one week and 6 months after completed intervention
  WAI is a questionnaire, which serves to conduct a self-assessment. The focus is on the employees and their work ability assessed by themselves
Change in Cough frequency | Change from baseline cough frequency at one week and 6 months after completed intervention
  24 hour consecutive recording of cough frequency in home environment
Change in the hypersensitivity of the cough reflex | Change from baseline hypersensitivity of the cough reflex at one week after completed intervention
  Standardised provocation test with inhaled hypertonic saline
Change in inflammation biomarkers in blood; eosinophil count | Change from baseline inflammation biomarkers (eosinophil count) in blood at one week after completed intervention
  Blood samples for eosinophil count, (cells/l)
Change in inflammation biomarker fractional exhaled nitric oxide (FeNO) | Change from baseline FeNo at one week after completed intervention
  Measured exhaled nitric oxide (NO) at 50 mL/s using a chemiluminescence NO analyzer.
Change in inflammation biomarkers in blood; level of eosinophil cationic protein (ECP) | Change from baseline inflammation biomarkers in blood (ECP) at one week after completed intervention
  Blood samples for ECP (mcg/l)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Wallstedt, Study Director — Uppsala Academical Hospital, Uppsala, Sweden
Locations (1):
- Uppsala Academical Hopsital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No